CLINICAL TRIAL: NCT03721380
Title: Efficacy of Drug and Risk Behavior Counseling Intervention Among Injecting Drug Users at Opioid Substitution Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University (Other)
Responsible Party: Principal Investigator, Tony Szu-Hsien Lee, Professor, National Taiwan University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: BDRC
Record Dates: First submitted 2018-10-23; First posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Substance Use Disorders
Keywords: Behavior drug and risk reduction counseling; Heroin; Addiction treatment; Randomization; Treatment effect
MeSH Terms: conditions — Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BDRC (Experimental): At the time of assignment to the counseling intervention arm of the study, there will be an initial meeting between the subject and the assigned counselor. As described in the counseling manual, this initial session is designed to introduce the counselor, review the purpose and expectations of counseling, review the rules of confidentiality, agree on attendance times and rescheduling rules, and to begin to collect information from the participant on their drug use and risk behaviors. Behavioral contracting is a key component to this counseling approach.
  Interventions: Behavioral: Treatment as usual
- TAU (Other): Patients receive some HIV risk education for the enrollment; after that, health education is delivered irregularly (1-2 times a month or none), based on the patient's needs.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Treatment as usual — Patients receive some HIV risk education for the enrollment; after that, health education is delivered irregularly (1-2 times a month or none), based on the patient's needs. During MMT treatment, the participant receives monthly random urine testing for opiate use and HIV testing as needed. Monthly meetings between the patient and physician are expected to occur however, there is no structure to these sessions and content is considered to be quite variable.
  Other Names: Methadone treatment with Bi-weekly counseling using BDRC

SUMMARY:
Behavior drug and risk reduction counseling (BDRC), a structured, non-intense, cognitive-behavioral approach intervention designed to increase methadone maintenance treatment retention and reduce drug use and related risk behaviors among IDUs.

DETAILED DESCRIPTION:
Techniques of the Cognitive Behavior Therapy combined with drug dependence psychoeducation was developed by research team. BDRC consists of 12 sessions, including an initial session, 3 drug education sesssions, psychosocial counseling and behavioral skills. This initial session is designed to introduce the counselor, review the purpose and expectations of counseling, review the rules of confidentiality, agree on attendance times and rescheduling rules, and to begin to collect information from the participant on their drug use and risk behaviors. Behavioral contracting is a key component to this counseling approach. Drug education focuses on how heroin may influence patients' cognitive function and their HIV/HCV risk behaviors. Counseling and behavior skills trained patients to reflect their thoughts and learned new life skills in order to delay or abstrain from heroin use.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in opioid substitution treatment
* Injected heroin within past 30 days by self-report, documented by "tracks" or puncture marks
* 20 or more years of age
* Meets ICD-10 criteria for opiates dependence with physiologic features
* Agrees to keep bi-weekly appointments if selected
* Current address within Taipei and Keelung, and not planning to move
* Willingness and ability to give informed consent and otherwise participate
* Provision of adequate locator information

Exclusion Criteria:

* Clinically significant cognitive impairment, schizophrenia, paranoid disorder, bipolar disorder
* Advanced neurological, cardiovascular, renal, or other medical disorder that is likely to impair or make hazardous patient's ability to participate
* Physiologically dependent on alcohol, benzodiazepines or other sedative type drugs
* Concurrent participation in another treatment study
* Planning to enter inpatient or residential treatment within next year
* Pending legal charges with likely incarceration within next 12 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2012-05-14 (Actual); Primary Completion 2014-07-31 (Actual); Study Completion 2015-07-31 (Actual)

PRIMARY OUTCOMES:
Change in heroin use | 3, 6, and 12 months
  Testing patients' urine for heroin use

SECONDARY OUTCOMES:
Number of treatment section | Within 6 months
  How many counseling sessions attended by patients?

CONTACTS AND LOCATIONS:
Overall Officials: Tony Szu-Hsien Tony Szu-Hsien, Ph.D., Principal Investigator — National Taiwan University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chawarski MC, Zhou W, Schottenfeld RS. Behavioral drug and HIV risk reduction counseling (BDRC) in MMT programs in Wuhan, China: a pilot randomized clinical trial. Drug Alcohol Depend. 2011 Jun 1;115(3):237-9. doi: 10.1016/j.drugalcdep.2010.09.024. Epub 2010 Dec 14. PMID 21159452
- See also: This pilot clinical trial evaluated whether the efficacy of methadone maintenance treatment (MMT) provided with limited psychosocial services is improved by the addition of manual-guided behavioral drug and HIV risk reduction counseling (BDRC). — http://www.ncbi.nlm.nih.gov/pubmed/?term=Behavioral+drug+and+HIV+risk+reduction+counseling+(BDRC)+in+MMT+programs+in+Wuhan%2C+China%3A+a+pilot+randomized+clinical+trial.